CLINICAL TRIAL: NCT07042659
Title: Effectiveness of an Accelerated Photobiomodulation Protocol With Blue Light in Patients With Hard-to-heal Wounds: a Single-arm Clinical Trial
Brief Title: Effectiveness of Blue Light for Hard-to-heal Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Blue_light_chronic_wounds
Record Dates: First submitted 2025-06-17; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Hard-to-heal Wounds; Chronic Wounds; Wound Healing Delayed; Photobiomodulation Therapy
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Photobiomodulation group (Experimental): Participants in the intervention group will receive an accelerated photobiomodulation protocol using a portable blue LED device (EmoLED™, 415 nm, 120 mW/cm², 7.2 J/cm²), applied twice weekly for 4 weeks in a nurse-led outpatient clinic. Each treatment is administered after wound bed preparation and in combination with standard wound care (cleansing, appropriate dressings, and compression therapy when indicated). Wound area, pain, exudate, and surrounding skin condition are assessed at baseline, at week 4, and at week 12 follow-up. No control arm is included.
  Interventions: Device: Photobiomodulation

INTERVENTIONS:
Device: Photobiomodulation — Accelerated photobiomodulation therapy using EmoLED™, a portable blue LED device (415 nm, 120 mW/cm², 7.2 J/cm²). The device delivers continuous blue light at 4 cm from the wound surface, 60 seconds per 25 cm² sub-area (120 seconds for diabetic wounds), administered twice weekly for 4 consecutive weeks. The protocol is combined with standard wound care (cleansing, dressings, compression as indicated). The intervention is designed to promote wound healing in hard-to-heal wounds by modulating inflammation, enhancing angiogenesis, fibroblast activation, and re-epithelialization. This accelerated protocol (twice weekly vs. standard weekly regimens) aims to optimize clinical outcomes in a nurse-led outpatient setting and distinguishes this intervention from lower-frequency or red/infrared-based photobiomodulation approaches.

SUMMARY:
Hard-to-heal wounds-those that fail to heal despite appropriate treatment-are a growing clinical challenge, often leading to significant discomfort, reduced quality of life, and high healthcare costs. These wounds are common among older adults and individuals with chronic conditions such as venous disease, diabetes, and lymphatic disorders. Photobiomodulation, a non-invasive therapy that uses specific wavelengths of light to stimulate biological processes, has shown promise in promoting wound healing. However, its effectiveness for long-standing, treatment-resistant wounds is not yet well established.

This pilot study aims to evaluate the effects of an accelerated photobiomodulation protocol using blue light in patients with hard-to-heal wounds. The study takes place in nurse-led outpatient wound care clinics within the local health authority of Turin (ASL Città di Torino, Italy), which serves a diverse urban population.

Eligible patients are adults with venous, diabetic, lymphatic, or mixed etiology wounds that have remained unhealed for at least two years. Participants receive blue light photobiomodulation treatment twice weekly for four weeks, in addition to standard wound care. Each session includes direct application of blue light to the wound area, following appropriate wound bed preparation and dressing changes.

The primary outcome is the reduction in wound size, measured at baseline, at the end of treatment (week 4), and at a follow-up visit (week 12). Secondary outcomes include changes in pain levels, wound exudate characteristics, and the condition of surrounding skin. Adverse events are monitored throughout the study.

By testing a standardized and replicable treatment protocol, this study seeks to generate preliminary evidence on whether blue light photobiomodulation can safely and effectively enhance healing in this complex patient population. Results may inform future clinical guidelines and support the integration of photobiomodulation into routine wound care pathways.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years;
* Presence of at least one hard-to-heal wound (defined as a wound unhealed despite treatment for ≥ 2 years);
* Wound etiology of venous, lymphatic, diabetic, or mixed origin (venous/lymphatic/arterial documented);
* Wound suitable for photobiomodulation treatment according to clinical evaluation;
* Ability to provide written informed consent;
* Willingness and ability to comply with the study protocol and attend scheduled visits.

Exclusion Criteria:

* Age < 18 years;
* Active oncological disease;
* Wound of exclusively arterial etiology;
* Wound with active infection at the time of enrollment;
* Participation in another interventional clinical trial within the past 3 months;
* Any medical or psychological condition that, in the investigator's judgment, would interfere with study participation or pose an unacceptable risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Wound Area Change | Baseline, Week 4 (end of treatment), Week 12 (follow-up)
  The primary outcome is the change in wound area (cm²) from baseline to week 12. Wound area is measured using CutiMed® Wound Navigator, a validated digital tool for wound assessment. The wound is photographed and measured at three timepoints: baseline, week 4 (end of photobiomodulation treatment), and week 12 (follow-up). The change in area is calculated as both absolute change (in cm²) and percentage change from the baseline. The outcome will assess the effectiveness of the accelerated photobiomodulation protocol in promoting long-term wound healing in patients with hard-to-heal wounds.

SECONDARY OUTCOMES:
Pain Change | Baseline, Week 4 (end of treatment), Week 12 (follow-up)
  Pain intensity reported by participants using a 0-10 Numeric Rating Scale (NRS). Pain is assessed at each treatment session, at the end of photobiomodulation treatment (week 4), and at week 12 follow-up. Change in pain score over time will be analyzed.
Change in Wound Exudate Quantity | Baseline, Week 4 (end of treatment), Week 12 (follow-up)
  Wound exudate quantity is assessed by nurses using a 4-point Likert scale (0 = absent; 1 = scarce; 2 = moderate; 3 = abundant). Assessed at each treatment session, at week 4, and at week 12 follow-up to monitor wound response to treatment.
Change in Wound Exudate Quality | Baseline, Week 4 (end of treatment), Week 12 (follow-up)
  Wound exudate quality is assessed by nurses using a 4-point Likert scale (0 = clear; 1 = slightly bloody; 2 = bloody; 3 = purulent). Assessed at each treatment session, at week 4, and at week 12 follow-up to evaluate wound progression and infection status.
Change in Surrounding Skin Condition | Baseline, Week 4 (end of treatment), Week 12 (follow-up)
  Condition of skin surrounding the wound is assessed by nurses using a 4-point Likert scale (0 = healthy pink; 1 = slightly reddened; 2 = reddened; 3 = inflamed). Assessed at each treatment session, at week 4, and at week 12 to monitor local inflammation and skin integrity.

CONTACTS AND LOCATIONS:
Overall Officials: Alessio Conti, PhD, Principal Investigator — ASL Citta di Torino
Locations (1):
- ASL Citta di Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: No
Given the small sample size and potential identifiability of individual cases, individual participant data will not be publicly shared. Aggregate data may be made available upon reasonable request to the corresponding author.